CLINICAL TRIAL: NCT03779932
Title: Generation of Prediction Equations to Analyze Body Composition of Obese Adults Based on Bioelectrical Impedance Analysis (BIA)
Brief Title: Generation of Prediction Equations to Analyze Body Composition of Obese Adults Based on BIA
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-20
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2018-12

CONDITIONS: Bioelectrical Impedance Measurement of Healthy Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was based on the clinical trial BCA-01 (NCT01368640) "Generation of prediction equations to analyze body composition of adults based on Bioelectrical Impedance Analysis (BIA)" and implicates an extension of the study collective. Aim of the study is to develop prediction equations for calculating FFM, TBW, ECW and SMM based on the gold standard reference methods ADP, DXA, MRI, D2O and NaBr on the one hand and measurement data of the BIA devices on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults in an
* age range of 18 to 65 years
* BMI > 30 kg/m2

Exclusion Criteria:

* acute and chronic diseases
* regular intake of medications (except for contraceptives)
* amputation of limbs
* electrical implant as cardiac pacemaker
* insulin pumps
* artificial joints
* metallic implants (except tooth implants)
* claustrophobia
* pregnancy or breastfeeding period
* probands who cannot provide an ICF by themselves
* probands who might be dependent from the sponsor or the inv. site
* current alcohol abuse
* frequent hypersensitivity reactions/allergies determ. anamnestically
* extensive tattoos at arms or legs

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 38 healthy obese adults
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2016-02-24 (Actual); Study Completion 2016-02-24 (Actual)

PRIMARY OUTCOMES:
BIA 5 and 50 kHz | 15 minutes
  Bioelectrical Impedance of 5 and 50 kHz for one body side
BIA 50 kHz | 15 minutes
  Bioelectrical Impedance of 50 kHz for all 4 extremities
Total body water | 15 minutes
  Total body water (TBW) by deuterium (D2O) dilution
Extracellular water | 15 minutes
  Extracellular water (ECW) by NaBr dilution
Fat-free mass | 1 hour
  Fat-free mass by a 4-compartment model based on dual energy x-ray absorption (DXA), air displacement plethysmography (ADP), D2O dilution and weight
Skeletal muscle mass | 1 hour
  Skeletal muscle mass (SMM) by magnetic resonance imaging (MRI)
Visceral adipose tissue | 1 hour
  Visceral adipose tissue VAT by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Complete BIA | 15 minutes
  Bioelectrical Impedance of 1, 1.5, 2, 3, 7.5, 10, 15, 20, 30, 75, 100, 150, 200, 300, 500, 750 and 1,000 kHz for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred J Müller, Prof. Dr., Principal Investigator — Christian-Albrechts-University of Kiel
Locations (1):
- Institute of Human Nutrition and Food Science, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Enderle J, Reljic D, Jensen B, Peine S, Zopf Y, Bosy-Westphal A. Normal values for body composition in adults are better represented by continuous reference ranges dependent on age and BMI. Clin Nutr. 2023 May;42(5):644-652. doi: 10.1016/j.clnu.2023.03.006. Epub 2023 Mar 9. PMID 36933351
- [Derived] Jensen B, Braun W, Both M, Gallagher D, Clark P, Gonzalez DL, Kluckmann K, Bosy-Westphal A. Configuration of bioelectrical impedance measurements affects results for phase angle. Med Eng Phys. 2020 Oct;84:10-15. doi: 10.1016/j.medengphy.2020.07.021. Epub 2020 Jul 30. PMID 32977906